CLINICAL TRIAL: NCT05937269
Title: Assessing Impact of Early Physiotherapy on Lymphatic Dysfunction in Head and Neck
Brief Title: Assessing Impact of Early Physiotherapy on Lymphatic Dysfunction in Head and Neck Cancer Survivorship
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, John Rasmussen, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-23-0268
Record Dates: First submitted 2023-06-22; First posted 2023-07-10 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Lymphedema of Face; Head and Neck Cancer
Keywords: indocyanine green imaging; head and neck cancer-acquired lymphedema; near-infrared fluorescence lymphatic imaging; advanced pneumatic compression therapy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Advanced Pneumatic Compression (Experimental): Subjects who present with dermal lymphatic backflow will be asked to complete a session of advanced pneumatic compression therapy each day at home.
  Interventions: Combination Product: Near-infrared fluorescence lymphatic imaging; Device: advanced pneumatic compression therapy
- Standard-of-Care (Active Comparator): Subjects who present with dermal lymphatic backflow will continue under standard-of-care surveillance of lymphedema and will only receive treatment if they are diagnosed with head and neck cancer-acquired lymphedema.
  Interventions: Combination Product: Near-infrared fluorescence lymphatic imaging
- No Dermal Backflow (Other): Subjects who do not present with dermal lymphatic backflow at enrollment will be monitored at subsequent visits and if/when dermal lymphatic backflow is observed will be randomized into either Advanced Pneumatic Compression or Standard-of-Care arm.
  Interventions: Combination Product: Near-infrared fluorescence lymphatic imaging

INTERVENTIONS:
Combination Product: Near-infrared fluorescence lymphatic imaging — All subjects will undergo lymphatic imaging at enrollment, 3, 6, and 12 months to assess the extent of dermal lymphatic backflow. Small amounts (0.1 mL) of a solution of indocyanine green (ICG) will be intradermally injected near the ear and along the jaw. Images of the lymphatics will be acquired by shining a dim light on the face and neck and acquiring the resulting fluorescent signal emanating from ICG-laden lymph. Images will be processed to calculate the area of the head and neck that show abnormal dermal lymphatic backflow.
  Other Names: indocyanine green imaging
Device: advanced pneumatic compression therapy — The advanced pneumatic compression device (APCD) mimics manual lymphatic drainage, a light massage that stimulates lymphatic uptake and function and frequently prescribed for lymphedema therapy.
  Arms: Advanced Pneumatic Compression

SUMMARY:
The goal of this clinical trial is to learn if treating the lymphatics in head and neck cancer survivors before clinical diagnosis of lymphedema will prevent its development or progression. The main questions it aims to answer are:

* Does early lymphatic treatment, before onset of clinical symptoms, prevent the development of head and neck lymphedema?
* Does dermal lymphatic backflow provide an early indication of lymphedema and its response to treatment?

Over the course of one year, participants will undergo several sessions near-infrared fluorescence lymphatic imaging to assess whether they have abnormal dermal lymphatic backflow following head and neck cancer treatment. Subjects will be divided into two groups, a treated and a control group. The treated group will be asked to complete daily sessions of pneumatic compression therapy at home, while the control group will receive standard-of-card treatment after clinical diagnosis of lymphedema. Researchers will compare the incidence of lymphedema between the two groups to see if treatment before diagnosis prevents the development and progression of head and neck lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years of age or older
* Participants must have previously been diagnosed with head and neck cancer and undergone surgery and radiation as part of their standard-of-care treatment plan
* Participants must be ≥ 4 weeks but less than 3 months post-radiation therapy at enrollment
* Female participants of childbearing potential must have a negative urine pregnancy test ≤ 36 hours prior to study drug administration
* Female participants of childbearing potential must agree to use a medically accepted method of contraception for a period of one month after each imaging session
* Male participants must agree to shave facial hair on imaging days
* Participants must be willing and able to independently use the pneumatic compression device at home daily for up to 12 months as directed by study personnel.

Exclusion Criteria:

* Persons who are pregnant or breast-feeding
* Females of child-bearing potential, who do not agree to use an approved contraceptive for one month after each imaging session
* Persons who do not meet inclusion criteria
* Iodine allergy
* Persons with a chest circumference of 150 cm or more
* Uncontrolled hyperthyroidism or parathyroidism (for which an endocrinologist recommends against neck compression)
* Carotid sinus hypersensitivity syndrome
* Symptomatic carotid artery disease, as manifested by a recent transient ischemic attack (within 30 days), ischemic stroke or amaurosis fugax (monocular visual ischemic symptoms or blindness)
* Symptomatic bradycardia in the absence of a pacemaker or internal jugular venous thrombosis (within 3 months)
* Increased intracranial pressure or other contraindication to internal or external jugular venous compression
* Acute radiation dermatitis, unhealed surgical scar, unhealed or open wound(s), surgical flap less than 6 to 8-weeks post-operative
* Facial or head and neck dermal metastasis
* Acute facial infection (e.g., facial, or parotid gland abscess)
* Heart failure (acute pulmonary edema, decompensated acute heart failure)
* Acute venous disease (acute thrombophlebitis, acute deep venous thrombosis, acute pulmonary embolism)
* Severe peripheral artery disease (critical limb ischemia including ischemic rest pain, arterial wounds, or gangrene)
* Active skin or limb infection/inflammatory disease (acute cellulitis, other uncontrolled skin, or untreated inflammatory skin disease)
* Any condition where increased venous and lymphatic return is undesirable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence/Severity of lymphedema | Enrollment
  The incidence of lymphedema between the control and treated groups will be compared.
Incidence/Severity of lymphedema | 3 months
  The incidence of lymphedema between the control and treated groups will be compared.
Incidence/Severity of lymphedema | 6 months
  The incidence of lymphedema between the control and treated groups will be compared.
Incidence/Severity of lymphedema | 12 months
  The incidence of lymphedema between the control and treated groups will be compared.

SECONDARY OUTCOMES:
Change in area of dermal lymphatic backflow | 3 months
  The change (from enrollment) in the area of the head and neck that is covered by abnormal dermal lymphatic backflow as assessed using near-infrared fluorescence lymphatic imaging.
Change in area of dermal lymphatic backflow | 6 months
  The change (from 3 months) in the area of the head and neck that is covered by abnormal dermal lymphatic backflow as assessed using near-infrared fluorescence lymphatic imaging.
Change in area of dermal lymphatic backflow | 12 months
  The change (from 6 months) in the area of the head and neck that is covered by abnormal dermal lymphatic backflow as assessed using near-infrared fluorescence lymphatic imaging.

CONTACTS AND LOCATIONS:
Overall Officials: John Rasmussen, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Results will be published in a scientific journal along with description of protocol. The complete data set includes large (GBs) sequences of images as well as protected health information (faces). Partial, redacted data sets may be sharable upon request.